CLINICAL TRIAL: NCT02705820
Title: A Phase II Study of Switch Maintenance Pembrolizumab in Patients With Non Small Cell Lung Cancer (NSCLC) Who do Not Progress After First Line Platinum Doublet Chemotherapy. (SWIPE)
Brief Title: Switch Maintenance Pembrolizumab in Patients With NSCLC After First Line Platinum Doublet Chemotherapy
Acronym: SWIPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bank of Cyprus Oncology Centre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Haris Charalambous, Dr Haris Charalambous BM MRCP FRCR, Bank of Cyprus Oncology Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-449
Record Dates: First submitted 2016-02-25; First posted 2016-03-11 (Estimated); Results first posted 2025-01-24 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Non Small Cell Lung Cancer
Keywords: Metastatic, Lung Cancer, Switch, Maintenance, Pembrolizumab.
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm study (Experimental): experimental treatment with maintenance pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Switch maintenance pembrolizumab treatment
  Other Names: MK-3475

SUMMARY:
Single arm one stage Phase II study: post 4-6 cycles platinum doublet chemotherapy for patients with metastatic Non Small Cell Lung Cancer (NSCLC) offering Pembrolizumab as maintenance therapy to non-progressors with primary endpoint: Immune Related Progression Free Survival (irPFS) at 1 year. Aim to show that this is at least 25% (compared to an expected 12% 1 year PFS based on the Pemetrexed and Erlotinib maintenance trials).

DETAILED DESCRIPTION:
Rationale:

There are currently no data on maintenance therapy with PD1/ PDL1 inhibitors in NSCLC. After an initial response / stable disease to first line chemotherapy, non-progressors / candidates for maintenance treatment, represent an ideal setting / patient group to test the efficacy of Pembrolizumab given that chemotherapy results in antigen release, hence it has the potential to augment immune checkpoint blockade, and following disease cytoreduction, this represents a lower disease burden setting, that may suit checkpoint inhibition better given the recent studies in Prostate cancer with Ipilimumab and Melanoma with Pembrolizumab(suggesting better outcomes for patients with less extensive disease).

Primary endpoint: percentage of patients that have not progressed at 1 year using immune related radiological criteria.

All patients to be treated with fixed dose 200mg iv Pembrolizumab until unacceptable toxicity, disease progression or completion of 2 years therapy.

Statistical Analysis Plan Summary The study employs a one stage phase II Fleming's design using irPFS at 1 year as primary endpoint. Using response hypotheses of H0 < 12 % and Ha> 25% i.e. that the irPFS at 1 year for the maintenance Pembrolizumab arm is 25%, compared to 12% in the normal chemotherapy maintenance arm, with a significance level (i.e., the probability of rejecting H0 when it is true) α=0.05 and the power (i.e. the probability of deciding the regimen is active) is 0.8 when true response rate is 25%, 48 patients are required to be entered into this study.

Entry Criteria Diagnosis/Condition for Entry into the Trial In order to be eligible for trial entry, patients must have a diagnosis of metastatic Non Small Cell Lung Cancer, and should not have progressed after first line palliative chemotherapy with a platinum doublet. They should have received no more than six (6) cycles of a platinum doublet chemotherapy, and should be able to receive treatment within three (3) to six (6) weeks from the last chemotherapy administration.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible for participation in this trial, the subject must:

  1. Be willing and able to provide written informed consent/assent for the trial.
  2. Be above 18 years of age on day of signing informed consent.
  3. Have measurable disease based on RECIST 1.1.
  4. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
  5. Have a performance status of 0 to 2 on the ECOG Performance Scale.
  6. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

     Table 1 Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Renal Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN, AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 g/L Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
  7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
  8. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

     Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
  9. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Have completed more than six (6) cycles of first line platinum doublet chemotherapy or more than six (6) have elapsed from the last chemotherapy administration of the first line chemotherapy with platinum doublet.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a known history of active TB (Bacillus Tuberculosis)
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Haris Charalambous, BM MRCP FRCR, Principal Investigator — Consultant Oncologist, BOC Oncology Centre
Locations (1):
- Bank of Cyprus Oncology Centre, Nicosia, Strovolos, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kakouri AC, Spiliotaki M, Loizidou EM, Stylianou I, Papageorgiou E, Panayi CG, Constantinou AI, Charalambous H, Deltas C, Papagregoriou G. Monitoring pembrolizumab response in patients with metastatic non-small cell lung cancer using circulating tumour DNA and circulating tumour cells. Transl Lung Cancer Res. 2025 Jun 30;14(6):1945-1960. doi: 10.21037/tlcr-2024-1095. Epub 2025 Jun 26. PMID 40673096
- [Derived] Charalambous H, Brown C, Vogazianos P, Katsaounou K, Nikolaou E, Stylianou I, Papageorgiou E, Vraxnos D, Aristodimou A, Chi J, Costeas P, Shammas C, Apidianakis Y, Antoniades A. Dysbiosis in the Gut Microbiome of Pembrolizumab-Treated Non-Small Lung Cancer Patients Compared to Healthy Controls Characterized Through Opportunistic Sampling. Thorac Cancer. 2025 May;16(9):e70075. doi: 10.1111/1759-7714.70075. PMID 40356191

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm Study
Started | 48
Completed | 9
Not Completed | 39
Not completed — Death | 2
Not completed — Disease Progression | 34
Not completed — Clinical Deterioration | 3

BASELINE CHARACTERISTICS:
Population: Pembrolizumab is administrated at 200 mg fixed dose i.v. on day 1 of every 3 week cycle for a maximum or 2 years (expected maximum of 36 doses), or until progression of disease determined according to immune related Response Criteria (irRC) or lack of tolerability, or until the patient declines further treatment for patients that have not progressed to first line chemotherapy for advanced / metastatic NSCLC.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 66 [40 to 82]
Age, Customized [Count of Participants; unit: Participants]
  <70 years | 30
  ≥70 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 47
  Asian | 1
Number of Participants [Number; unit: participant] — Patients with metastatic NSCLC who have not progressed after first line chemotherapy, were identified by the treating oncologists and enrolled as per eligibility criteria.
  participant | 48

OUTCOME MEASURES:

1. Primary Outcome: Immune Related Progression Free Survival (irPFS) at 1 Year
Description: To investigate whether treatment with pembrolizumab improves 1 year irPFS, compared to historical controls (from the Pemetrexed and Erlotinib maintenance trials). Aim to show that this is at least 25% (compared to an expected 12% 1 year PFS based on the Pemetrexed and Erlotinib maintenance trials) using a one stage phase II Fleming's design.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 48
Participants | 16

2. Secondary Outcome: Response Rates Using RECIST Version 1.1
Description: Response rates according to RECIST criteria Version 1.1 where Complete response(CR): Disappearance of all target lesions. Partial response(PR): At least a 30% decrease in the sum of diameters of all target lesions, (from baseline sum of diameters in the absence of CR). Progressive disease(PD): Any new lesion or at least a 20% increase in the sum of diameters of target lesions, (from the smallest sum of diameters at prior timepoints -including baseline). Stable disease(SD): Neither CR or a PR nor sufficient increase to qualify for PD.
Time Frame: 7 years
Population: In order to be eligible for trial entry, patients must have a diagnosis of metastatic Non Small Cell Lung Cancer, and should not have progressed after first line palliative chemotherapy with a platinum doublet. They should have received no more than six (6) cycles of a platinum doublet chemotherapy, and should be able to receive treatment within three (3) to six (6) weeks from the last chemotherapy administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 48
Participants
  Complete Response | 1
  Partial Response | 6
  Non- Responders | 41

3. Secondary Outcome: Response Rates With Immune Related Response Criteria (irRC)
Description: Response rates according to RECIST criteria. Time from randomization of the first patient until database cut-off date for the final analysis (Jul 2016 - May 2023; approximately 7 years).
Time Frame: 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 48
Participants
  Complete Response | 1
  Partial Response | 6
  Non Responders | 41

4. Secondary Outcome: Radiological Progression Free Survival (PFS) Using RECIST Criteria Version 1.1
Description: PFS calculated using RECIST criteria. RECIST Criteria Version 1.1: Complete response(CR): Disappearance of all target lesions. Partial response(PR): At least a 30% decrease in the sum of diameters of all target lesions, (from baseline sum of diameters in the absence of CR). Progressive disease(PD): Any new lesion or at least a 20% increase in the sum of diameters of target lesions, (from the smallest sum of diameters at prior timepoints -including baseline). Stable disease(SD): Neither CR or a PR nor sufficient increase to qualify for PD. Immune related irPFS calculated using Immune related Response criteria where upon PD there a CT scan would be repeated in 4-6 weeks to exclude pseudoprogression..
Time Frame: 7 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm Study
Number analyzed (Participants) | 48
months | 2.1 [0.0 to 4.2]

5. Secondary Outcome: Immune-related PFS Using irRC
Description: PFS calculated using RECIST criteria. Immune related irPFS calculated using Immune related Response criteria.
Time Frame: 7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm Study
Number analyzed (Participants) | 48
months | 6.3 [4.2 to 8.4]

6. Secondary Outcome: Overall Survival
Description: Defined as time from the date of randomisation until death from any cause or time to the last follow up appointment (censored).
Time Frame: 7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm Study
Number analyzed (Participants) | 48
months | 12.2 [7.8 to 16.6]

7. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Assessed through analysis of the worst grade of toxicity/adverse events according to CTCAE v4.0 criteria observed over the whole treatment period. Adverse events are collected from study treatment initiation to 30 days after treatment is ceased for any reason. Serious adverse events and events of clinical interest are collected within 90 days after last dose of trial treatment.
Time Frame: 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 48
Participants
  Experienced any adverse event (any grade) | 48
  Experienced treatment related adverse event (any grade) | 42
  Experienced treatment related adverse event of grade 3-5 | 11

ADVERSE EVENTS:
Time Frame: Time from randomization of the first patient until database cut-off date for the OS analysis (Jul 2016 - May 2023; approximately 7 years).
Description: In the 'All-Cause Mortality' and the 'Serious Adverse Events' and 'Other (Not Including Serious) Adverse Events' sections, number of at risk patients includes all randomized patients, as all patients received at least one dose of trial treatment.
Arm/Group | Single Arm Study
All-Cause Mortality (participants affected / at risk) | 42/48
Serious Adverse Events (participants affected / at risk) | 13/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Study (N=48)
Hypotension (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Adrenal Insufficiency (Endocrine disorders) | 1
Hyperglycaemia (Endocrine disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Infections and Infestations (Infections and infestations) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Left Hip Fracture (Musculoskeletal and connective tissue disorders) | 1
Weakness of lower limb (Musculoskeletal and connective tissue disorders) | 1
Brachial Plexopathy (Nervous system disorders) | 1
Multi organ failure (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Study (N=48)
Platelet count decreased (Blood and lymphatic system disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 9
Non-Cardiac chest Pain (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Hypothyroism (Endocrine disorders) | 6
Hyperthyroism (Endocrine disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Gastroesophageal Reflux (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 21
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Nausea/dizziness (Gastrointestinal disorders) | 9
Pain (General disorders) | 12
Malaise (General disorders) | 26
Lung Infections (Infections and infestations) | 8
Bronchial Infection (Infections and infestations) | 6
Urinary Tract infection (Infections and infestations) | 2
Otitis external (Infections and infestations) | 2
Infection NOS (Infections and infestations) | 1
Gum Infection (Infections and infestations) | 1
Upper Respiratory Infection (Infections and infestations) | 4
Herpes Zoster (Infections and infestations) | 1
Fungus Infection (Infections and infestations) | 2
Non -neutropenic infection (Infections and infestations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Dysgeusia (Metabolism and nutrition disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 25
Alanine Transaminase (ALT) (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Weight Loss (Metabolism and nutrition disorders) | 13
Hyponatremia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 27
Neuralgia (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Fracture (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness of lower limbs (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensor neuropathy (Musculoskeletal and connective tissue disorders) | 1
Dysarthria (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 5
Anxiety (Psychiatric disorders) | 2
Creatinine increase (Renal and urinary disorders) | 2
Cystitis Noninfectious (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Urinary Frequency (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Flu like Syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial Stricture (Respiratory, thoracic and mediastinal disorders) | 4
Telangiectasias (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 17
Skin and Subcutaneous tissue disorders: other (Skin and subcutaneous tissue disorders) | 3
Rash maculopapular (Skin and subcutaneous tissue disorders) | 8
Superficial Thrombophlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT02705820/Prot_SAP_000.pdf